CLINICAL TRIAL: NCT05743231
Title: Comparison of Interpectoral Area Block+Serratus Anterior Area Block With Erector Spinae Block in Minimally Invasive Cardiac Surgery, Effect on Postoperative Pain and Recovery; Randomized Clinical Study
Brief Title: Comparison of Interpectoral+Serratus Anterior Block With Erector Spinae Block in Minimally Invasive Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Ayhan ŞAHİN, assistant professor, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022.212.11.13
Record Dates: First submitted 2023-01-13; First posted 2023-02-24 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pain
Keywords: pain management; regional anesthesia; minimally invasive cardiac surgery
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants will be randomly divided into two groups. The physician who will collect data in the cardiac surgery intensive care unit and cardiac surgery clinic will not know which group the participant is in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- interpectoral area block + serratus anterior area block group (IPSA) (Active Comparator): Interpectoral plane block + serratus anterior plane block will be performed randomly on the participants.
  Interventions: Procedure: interpectoral area block + serratus anterior area block group
- erector spinae group (ES) (Active Comparator): Erector spinae block will be performed randomly on the participants
  Interventions: Procedure: interpectoral area block + serratus anterior area block group

INTERVENTIONS:
Procedure: interpectoral area block + serratus anterior area block group — The interpectoral and serratus anterior area blocks will be applied immediately after general anesthesia is given to the participants under ultrasound guidance. 30 ml of 0.25% bupivacaine will be used for two blocks.
  Other Names: IPSA

SUMMARY:
Adequate pain management after minimally invasive cardiac surgery is essential for early ambulation and patient satisfaction. However, an incision similar to thoracotomy surgery is made by entering between the ribs, and a severely painful postoperative period is experienced as the intercostal nerves are cut.

Invasive cardiac surgery is necessary surgery that can take steps to improve the quality of life and functional status of patients without sternotomy. However, patients may experience intense pain in the immediate postoperative period, which can lead to inactivity, increased risk of complications, and greater consumption of opioids, resulting in adverse effects and prolonged hospital stays. Pain management is challenging due to a large number of dermatomes covered.

Interpectoral plane block + serratus anterior plane block, defined in 2012, has been used in many studies before as part of multimodal analgesia in minimally invasive cardiac surgery. Erector spinae block was also described in 2018 with positive results, which has been used in both sternotomies (open heart surgery) and minimally invasive procedures. Minimally invasive cardiac surgery can be excruciating in the postoperative period, just like thoracotomy surgeries. What is aimed in this study is to compare two previously known regional anesthesia techniques in this study.

DETAILED DESCRIPTION:
Minimally invasive cardiac surgery is necessary surgery that can take steps to improve the quality of life and functional status of patients without sternotomy. However, patients may experience intense pain in the immediate postoperative period, which can lead to inactivity, increased risk of complications, and greater consumption of opioids, resulting in adverse effects and prolonged hospital stays. Pain management is challenging due to a large number of dermatomes covered.

The interpectoral plane block + serratus anterior plane block seems to cover the thoracic dermatomes. It has been the subject of many studies in the same surgical group. Minimally invasive cardiac surgery can be excruciating in the postoperative period, just like thoracotomy surgeries. What is aimed of this study is to compare it with erector spinae block in this study. Additional anesthetic techniques, such as peripheral nerve blocks, are part of the multimodal analgesic strategy and are often used to manage acute pain better. Inadequate treatment can lead to persistent pain conditions. Although numerous nerve blocks exist for this purpose, some may fail because they do not cover the thoracic dermatomes or their entire innervation. The central hypothesis of this study hypothesis, interpectoral plane block + serratus anterior plane block, defined in 2012, has been used in many previous studies as part of multimodal analgesia in minimally invasive cardiac surgery. Erector spinae block was also described in 2018 with positive results that have been used in both sternotomies (open heart surgery) and minimally invasive procedures. In this randomized clinical trial, the study aims to compare the efficacy of previously known field blocks as part of multimodal analgesia in minimally invasive cardiac surgery. As presented in the literature, these techniques have been routinely performed so much that review articles have been written. Targeted in this study, preliminary results will be postoperative pain scores. At Namık Kemal University anesthesia clinic, It is regularly used as part of multimodal analgesia and resident training. Traditional intravenous analgesia methods cause many undesirable side effects depending on the type of opioid used, and they are insufficient compared to regional anesthesia methods.

The main aim of this study is to investigate the effectiveness of these two methods, routinely used in thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo cardiac surgery for the first time
* ASA I-III (American Society of Anesthesiology classification) patients between the ages of 18-75
* Patients with an average bleeding profile
* Patients who gave written consent to participate in the study
* Patients without local anesthetic allergy and a history
* Patients who have the intellectual level to use the patient-controlled analgesia device

Exclusion Criteria:

* Patients who have undergone open heart surgery before undergoing valve replacement and revision
* Patients who did not agree to participate in the study
* Patients with cancer primarily
* Patients with local anesthetic allergy and a history
* Patients who do not have the intellectual level to use a patient-controlled analgesia device
* Patients with abnormal bleeding profile
* Patients who were re-operated due to any surgical complication (bleeding, etc.) within the 24th hour after the operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) Pain Score at 24 Hours | 24 hours after surgery, following extubation
  A numerical ratio scale (NRS) requires the patient to rate pain on a defined scale. ifor example,0-10 where 0 is no pain and 10 is the worst pain imaginable.

SECONDARY OUTCOMES:
opioid consumption | up to 48 hours
  Patient-controlled analgesia (PCA) is a method of pain control that gives patients the power to control their pain. In PCA, a computerized pump called the patient-controlled analgesia pump, which contains a syringe of pain medication as prescribed by a doctor, is connected directly to a patient's intravenous (IV) line. (micrograms)
recovery criteria | up to 48 hours
  Postoperative recovery is an energy-requiring process that has four dimensions - physiological, psychological, social, and habitual recovery. The meaning after minimally invasive cardiac surgery; covers the parameters followed by the patient in the intensive care process and in the clinic. extubation time (from the moment of arrival in the intensive care unit/hr. Postoperative carbon dioxide levels in mmHg.Drainage amount in milliliters.
intraoperative | up to 48 hours
  As it is known, single-lung ventilation is performed in these patients until they enter the heart-lung pump. In the meantime, it is essential to determine whether there are changes in the NIRS( near-infrared spectroscopy monitor) values compared to the baseline in these cases.(%)
CPOT score until extubation | up to extubation time.
  Critical Care Pain Observation Tool (CPOT)The CPOT was developed for the assessment of pain in critically ill patients. The scale consists of four behavioral domains: facial expression, body movements, muscle tension and compliance with the ventilation for intubated patients.(0 to 8)
NRS at 6, 12, and 48 hours | From surgery to 6 hours, 12 hours, and 48 hours postoperatively
  Pain intensity was assessed at 6, 12, and 48 hours postoperatively using the 0-10 NRS scale, where 0 indicates no pain and 10 the worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- Namık Kemal University, Tekirdağ, Süleymanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No